CLINICAL TRIAL: NCT07148804
Title: Oral α-Amylase Enzyme Replacement for the Treatment of Diabetic Polyneuropathy
Brief Title: A Double-Blind, Placebo-Controlled Study of Fermented Deglycyrrhizinated Licorice Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mahmoud I Mostafa, Lecturer of Clinical Pharmacy, Faculty of Pharmacy, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6016A
Record Dates: First submitted 2025-08-11; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Polyneuropathy
Keywords: Diabetic complications; Diabetic polyneuropathy; Amylase deficiency; Licorice; FDGL
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented Deglycyrrhizinated Licorice (Active Comparator): Oral capsules containing 500 mg of fermented deglycyrrhizinated licorice root extract standardized to 2500 IU/gm of α-amylase enzyme and naturally occurring flavonoids and acid-lipase. Administered twice daily (1000 mg/day).
  Interventions: Drug: Fermented Deglycyrrhizinated Licorice
- Placebo Comparator (Placebo Comparator): 500 mg non-fermented deglycyrrhizinated licorice root extract capsules, matching FDGL in appearance, color, weight, and excipients. Administered twice daily.
  Interventions: Dietary Supplement: Non-fermented Deglycyrrhizinated Licorice

INTERVENTIONS:
Drug: Fermented Deglycyrrhizinated Licorice — Oral capsules containing 500 mg of fermented deglycyrrhizinated licorice root extract standardized to 2500 IU/gm of α-amylase enzyme and naturally occurring flavonoids and acid-lipase. Administered twice daily (1000 mg/day).
  Arms: Fermented Deglycyrrhizinated Licorice
Dietary Supplement: Non-fermented Deglycyrrhizinated Licorice — 500 mg non-fermented deglycyrrhizinated licorice root extract capsules, matching FDGL in appearance, color, weight, and excipients. Administered twice daily.
  Arms: Placebo Comparator

SUMMARY:
This double-blind, placebo-controlled study evaluated the efficacy of oral α-amylase enzyme replacement therapy in treating early-stage diabetic polyneuropathy (DPN). The study was conducted at Al-Azhar University Hospitals with 83 diabetic patients randomized to receive either fermented deglycyrrhizinated licorice extract (FDGL) containing α-amylase enzyme (2500 IU/gm) or placebo for 6 months. Primary outcomes measured improvements in nerve conduction velocity and vibration perception threshold.

DETAILED DESCRIPTION:
Diabetes mellitus complications continue to develop despite optimal glycemic control with insulin. Recent studies suggest that serum amylase deficiency correlates with the severity of diabetic complications. This study hypothesizes that α-amylase enzyme deficiency represents an enzymatic defect in the cascade between activated insulin receptors and mitochondrial energy liberation, contributing to diabetic complications.

α-amylase is a glycolytic enzyme that undergoes entero-pancreatic circulation and is proposed to be a precursor to key phosphorylating enzymes (glycogen phosphorylase, glucokinase, and hexokinase) essential for glycolysis. Supplementation with α-amylase may restore normal carbohydrate metabolism and prevent diabetic complications.

The study drug is a formulation rich in α-amylase enzyme prepared from fermented deglycyrrhizinated licorice root extract, also containing acid-lipase enzyme and naturally occurring flavonoids. The intervention was administered as 500mg capsules twice daily, one hour before meals, for 6 months alongside regular antidiabetic medications.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Type 1 or Type 2 diabetes mellitus
* Age between 15 and 65 years
* Diabetes duration of 1-5 years
* Body Mass Index (BMI) < 30 kg/m²
* HbA1c < 9%
* Serum creatinine < 2mg/dL
* Serum α-amylase < 45 IU/L (reference range: 28-100 IU/L)
* Vibration Perception Threshold (VPT) > 15V
* Absence of clinical symptoms of diabetic polyneuropathy

Exclusion Criteria:

* Treatment with medications that might influence nerve function (antiepileptic agents, tricyclic antidepressants, sympathomimetic agents)
* Presence of myopathies
* Presence of neuropathies from other causes
* Presence of malignancies
* Clinical symptoms of diabetic polyneuropathy
* Inability to comply with study protocol

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Sensory Nerve Conduction Velocity (SCV) | Baseline, 3 months, 6 months
  Measurement of nerve conduction velocity in sural nerve using digital electromyography equipment

SECONDARY OUTCOMES:
Motor Nerve Conduction Velocity (MCV) | Baseline, 3 months, 6 months
  Measurement of nerve conduction velocity in peroneal nerve using digital electromyography equipment
Vibration Perception Threshold (VPT) | Baseline, 3 months, 6 months
  Measurement using biothesiometer at six points on each foot (big toe, metatarsal bases, instep, heel)
Serum α-amylase Levels | Baseline, 3 months, 6 months
  Measurement of serum α-amylase concentration as marker of compliance and drug efficacy
Sensory Nerve Action Potential Amplitude (SNAP) | Baseline, 3 months, 6 months
  Amplitude measurement in sural nerve
Compound Muscle Action Potential Amplitude (CMAP) | Baseline, 3 months, 6 months
  Amplitude measurement in peroneal nerve

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aly Massoud, PhD, Study Chair — Department of Hepato-gastroenterology and Infectious Diseases, Faculty of Medicine, Al-Azhar University, Cairo, Egypt
Locations (1):
- Al-Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No